CLINICAL TRIAL: NCT02915523
Title: A Randomized, Placebo-controlled, Double-blind, Multicenter Phase 1b/2 Study of Avelumab With or Without Entinostat in Patients With Advanced Epithelial Ovarian Cancer Which Has Progressed or Recurred After First-line Platinum-based Chemotherapy and at Least Two Subsequent Lines of Treatment With a Safety Lead-in
Brief Title: Study of Avelumab With or Without Entinostat in Participants With Advanced Epithelial Ovarian Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Syndax Pharmaceuticals (Industry)
Collaborators: Merck KGaA, Darmstadt, Germany (Industry); Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SNDX-275-0603
Record Dates: First submitted 2016-09-14; First posted 2016-09-27 (Estimated); Results first posted 2024-01-10 (Actual); Last update posted 2024-01-10 (Actual); Status verified 2023-12

CONDITIONS: Epithelial Ovarian Cancer; Peritoneal Cancer; Fallopian Tube Cancer
Keywords: Ovarian Cancer; Histone Deacetylase Inhibitors; Entinostat; Solid tumor; Avelumab; SNDX-275; Ovarian Neoplasms; Ovarian Diseases; Fallopian Tube Cancer; Peritoneal Cancer
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial; Fallopian Tube Neoplasms; Ovarian Neoplasms; Ovarian Diseases | interventions — entinostat; avelumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Entinostat plus Avelumab (Active Comparator): Avelumab is administered intravenously (IV) on Day 1 of each 14-day cycle in combination with Entinostat administration on Day 1 and Day 8 of each cycle at the Maximum tolerated Dose (MTD)/RP2D as determined in the Phase Ib (Dose Determination) part of the study.
  Interventions: Drug: entinostat; Drug: avelumab
- Placebo plus Avelumab (Placebo Comparator): Avelumab is administered intravenously (IV) on Day 1 of each 14-day cycle in combination with placebo administered on Day 1 and Day 8 of each cycle.
  Interventions: Drug: avelumab; Drug: Placebo

INTERVENTIONS:
Drug: entinostat — An orally available histone deacetylases inhibitor (HDACi).
  Other Names: SNDX-275; MS-275
  Arms: Entinostat plus Avelumab
Drug: avelumab — A fully human antibody of the immunoglobulin (Ig) G1 isotype that targets and blocks Programmed death-ligand 1 (PD-L1), the ligand for Programmed cell death protein 1 (PD-1) receptor.
  Other Names: MSB0010718C
Drug: Placebo — A pill containing no active drug ingredient.
  Arms: Placebo plus Avelumab

SUMMARY:
The purpose of this study is to determine the biologically active dose of entinostat, when given in combination with avelumab, that is safe and warrants further investigation. Additionally, this study will evaluate the effectiveness of entinostat in combination with avelumab at the determined dose in terms of progression free survival compared to avelumab plus placebo in participants with refractory or recurrent epithelial ovarian cancer.

DETAILED DESCRIPTION:
The study is comprised of 2 phases: an open-label Safety Lead-in (Phase 1b) followed by an Expansion Phase (Phase 2). The Expansion Phase will evaluate the efficacy and safety of entinostat with avelumab when administered at the Recommended Phase 2 Dose (RP2D) versus avelumab alone in participants with advanced epithelial ovarian cancer in a randomized, double-blind, placebo-controlled setting. In Phase 2, participants will be randomized in a 2:1 ratio to receive avelumab plus entinostat or avelumab plus placebo, respectively.

All participants will be assessed at Screening and at specified times during the conduct of the study using standard clinical and laboratory assessments. Participants will be assessed for response through radiological assessments. Participants will continue receiving their appropriate cycles of study treatment until tumor progression or adverse events (AEs) occur which necessitate discontinuing therapy as determined by the Investigator.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed epithelial ovarian, fallopian tube, or peritoneal cancer
* Recurrent or progressive disease on or after initial platinum-based chemotherapy
* Evidence of measurable disease based on imaging studies within 28 days before the first dose of study drug
* Previously received at least 3, but no more than 6, lines of therapy including at least 1 course of platinum-based therapy
* Participant must have acceptable, applicable laboratory requirements
* Participants may have a history of brain metastasis provided certain protocol criteria are met
* Experienced resolution of toxic effect(s) of the most recent prior anti-cancer therapy to Grade ≤1 (except alopecia or neuropathy)
* Able to understand and give written informed consent and comply with study procedures.

Exclusion Criteria:

* Non-epithelial ovarian carcinomas or ovarian tumors with low malignant potential (i.e., borderline tumors)
* Another known malignancy that is progressing or requires active treatment (excluding adequately treated basal cell carcinoma or cervical intraepithelial neoplasia/cervical carcinoma in situ or melanoma in situ). Prior history of other cancer is allowed, as long as there is no active disease within the prior 5 years.
* Diagnosis of immunodeficiency or receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to enrollment.
* Active autoimmune disease that might deteriorate when receiving an immunostimulatory agent
* Previously treated with a histone deacetylase inhibitor (i.e., vorinostat, belinostat, romidepsin, panobinostat), PD-1/PD-L1-blocking antibody (i.e., atezolizumab, nivolumab, pembrolizumab), or a cytotoxic T-lymphocyte associated protein-4 (CTLA-4) agent
* Currently enrolled in (or completed) another investigational drug study within 30 days prior to study drug administration
* A medical condition that precludes adequate study treatment or increases participant risk

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2016-12-19 (Actual); Primary Completion 2019-02-21 (Actual); Study Completion 2021-04-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Meyers, MD, PhD, Study Director — Syndax Pharmaceuticals; Ursula Matulonis, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (12):
- United States (12):
  - H. Lee Moffitt Cancer Center and Research, Tampa, Florida
  - Florida Cancer Specialist East Region (SCRI Affiliate), West Palm Beach, Florida
  - University of Chicago, Chicago, Illinois
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins University, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - HCA Midwest Health (SCRI Affiliate), Kansas City, Missouri
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - University of Virginia, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: No
An independent data safety monitoring board (DSMB) will be established for the Phase 2 portion of this study to act in an advisory capacity to the Sponsor with respect to safeguarding the interests of trial patients and assessing the safety of the interventions administered during the trial.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study comprised 2 phases: an open-label Safety Lead-in (Phase 1b) and an Expansion Phase (Phase 2). Eligible participants were enrolled into Phase 1b or randomized into Phase 2 of the study within 3 days prior to starting study treatment on Cycle 1, Day 1.
Groups:
- Phase 1B: Avelumab + Entinostat (3 mg): Participants received entinostat 3 mg administered orally weekly (Days 1 and 8 of each 14-day cycle) in combination with avelumab intravenously (IV) once every 2 weeks (Day 1 of each 14-day cycle).
- Phase 1B: Avelumab + Entinostat (5 mg): Participants received entinostat 5 mg administered orally weekly (Days 1 and 8 of each 14-day cycle) in combination with avelumab IV once every 2 weeks (Day 1 of each 14-day cycle).
- Phase 2: Avelumab + Placebo: Participants received placebo matched to entinostat administered orally weekly (Days 1 and 8 of each 14-day cycle) in combination with avelumab IV once every 2 weeks (Day 1 of each 14-day cycle).
- Phase 2: Avelumab + Entinostat: Participants received entinostat at the maximum tolerated dose (MTD)/recommended Phase 2 dose (RP2D) (as determined in the Phase IB part of the study) administered orally weekly (Days 1 and 8 of each 14-day cycle) in combination with avelumab IV once every 2 weeks (Day 1 of each 14-day cycle).
Period: Dose Determination Phase (Phase 1B)
Arm/Group | Phase 1B: Avelumab + Entinostat (3 mg) | Phase 1B: Avelumab + Entinostat (5 mg) | Phase 2: Avelumab + Placebo | Phase 2: Avelumab + Entinostat
Started | 6 | 8 | 0 | 0
Received At Least 1 Dose Of Study Drug | 6 | 8 | 0 | 0
Dose-limiting Toxicity (DLT) Evaluable (Participants who received at least one dose of entinostat or avelumab were evaluated for DLTs over 2 cycles (Cycle 1 and Cycle 2).) | 6 | 8 | 0 (DLTs were not evaluated in Phase 2.) | 0 (DLTs were not evaluated in Phase 2.)
Completed | 0 | 0 | 0 | 0
Not Completed | 6 | 8 | 0 | 0
Not completed — Death | 5 | 4 | 0 | 0
Not completed — Sponsor Decision | 1 | 3 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0
Period: Expansion Phase (Phase 2)
Arm/Group | Phase 1B: Avelumab + Entinostat (3 mg) | Phase 1B: Avelumab + Entinostat (5 mg) | Phase 2: Avelumab + Placebo | Phase 2: Avelumab + Entinostat
Started | 0 | 0 | 41 | 85
Received At Least 1 Dose Of Study Drug | 0 | 0 | 40 | 85
Completed | 0 | 0 | 5 | 0
Not Completed | 0 | 0 | 36 | 85
Not completed — Death | 0 | 0 | 26 | 53
Not completed — Sponsor Decision | 0 | 0 | 4 | 22
Not completed — Withdrawal by Subject | 0 | 0 | 6 | 8
Not completed — Lost to Follow-up | 0 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Population: All participants who were enrolled in Phase 1B and randomized in Phase 2.
Groups:
- Phase 1B: Avelumab + Entinostat (3 mg): Participants received entinostat 3 mg administered orally weekly (Days 1 and 8 of each 14-day cycle) in combination with avelumab IV once every 2 weeks (Day 1 of each 14-day cycle).
- Phase 2: Avelumab + Entinostat: Participants received entinostat at the MTD/ RP2D (as determined in the Phase IB part of the study) administered orally weekly (Days 1 and 8 of each 14-day cycle) in combination with avelumab IV once every 2 weeks (Day 1 of each 14-day cycle).
- Total: Total of all reporting groups
Arm/Group | Phase 1B: Avelumab + Entinostat (3 mg) | Phase 1B: Avelumab + Entinostat (5 mg) | Phase 2: Avelumab + Placebo | Phase 2: Avelumab + Entinostat | Total
Number analyzed (Participants) | 6 | 8 | 41 | 85 | 140
Age, Customized [Count of Participants; unit: Participants]
  <65 years | 3 | 3 | 22 | 45 | 73
  ≥65 years | 3 | 5 | 19 | 40 | 67
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 8 | 41 | 85 | 140
  Male | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 2 | 2 | 4
  Not Hispanic or Latino | 6 | 8 | 37 | 80 | 131
  Unknown or Not Reported | 0 | 0 | 2 | 3 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 4 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 0 | 1
  Black or African American | 0 | 0 | 1 | 2 | 3
  White | 6 | 8 | 37 | 79 | 130
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Phase 2: Progression Free Survival (PFS), as Determined by the Local Investigator Using Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1)
Description: PFS was defined as the number of months from randomization to progressive disease (PD) or death due to any cause, whichever occurred first. PD: At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 millimeters (mm); the appearance of one or more new lesions; and unequivocal progression of existing non-target lesions.
Time Frame: From date of randomization to PD or death due to any cause (maximum exposure: 24 cycles [each cycle = 14 days])
Population: Full Analysis Set (FAS) included all participants who were randomized in Phase 2 by following the intent-to-treat principle.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 2: Avelumab + Placebo | Phase 2: Avelumab + Entinostat
Number analyzed (Participants) | 41 | 85
months | 1.51 [1.45 to 2.50] | 1.64 [1.41 to 2.69]
Statistical Analysis 1: Comparison: Phase 2: Avelumab + Placebo vs Phase 2: Avelumab + Entinostat; Test type: Other; Hazard Ratio (HR) = 0.899, 95% CI 2-sided [0.581 to 1.393] — Stratified HR estimated from a stratified univeriate Cox proportional hazards model. Avelumab + placebo was the reference treatment group

2. Primary Outcome: Phase 1b: Number of Participants With at Least One Dose Limiting Toxicity (DLT) Adverse Event (AE)
Description: A DLT was defined as the occurrence of any protocol-specified event within the first 2 cycles of treatment (from Cycle 1 Day 1 through the end of Cycle 2) of entinostat in combination with avelumab that were considered by the investigator to be at least possibly related to study drug.
Time Frame: Day 1 through Day 28 (Cycles 1 and 2)
Population: Safety analysis set included all participants who received at least 1 dose of either study drug, entinostat, or avelumab.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1B: Avelumab + Entinostat (3 mg) | Phase 1B: Avelumab + Entinostat (5 mg)
Number analyzed (Participants) | 6 | 8
Participants | 0 | 1

3. Secondary Outcome: Phase 1b: Recommended Phase 2 Dose (RP2D)
Description: The RP2D was determined in discussion with the Sponsor, Medical Monitor, and Dose Determination Phase Investigators. Additionally, observations related to immune correlates, and any cumulative toxicity observed after multiple cycles might be included in the rationale supporting the RP2D. The RP2D could be equal to or less than the preliminary maximum tolerated dose (MTD). The MTD was defined as the highest dose level at which <33% of 6 participants experienced DLT.
Time Frame: Day 1 through Day 28 (Cycles 1 and 2)
Population: as for outcome 2
Measure: Number; unit: mg
Groups:
- Phase 1B: Avelumab + Entinostat: Participants received entinostat 3 mg or 5 mg administered orally weekly (Days 1 and 8 of each 14-day cycle) in combination with avelumab IV once every 2 weeks (Day 1 of each 14-day cycle).
Arm/Group | Phase 1B: Avelumab + Entinostat
Number analyzed (Participants) | 14
mg | 5

4. Secondary Outcome: Phase 2: PFS, as Determined by the Local Investigator Using Immune Response RECIST (irRECIST)
Description: PFS was defined as the number of months from randomization to PD or death due to any cause, whichever occurred first. PD: Sum of the diameters (longest for non-nodal lesions, shortest for nodal lesions) of target and new measurable lesions increases ≥20% (compared to nadir), confirmed by a repeat, consecutive observation at least 4 weeks from the date first documented.
Time Frame: From date of randomization to PD or death due to any cause (maximum exposure: 24 cycles [each cycle = 14 days])
Population: FAS included all participants who were randomized in Phase 2 by following the intent-to-treat principle.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 2: Avelumab + Placebo | Phase 2: Avelumab + Entinostat
Number analyzed (Participants) | 41 | 85
months | 2.10 [1.45 to 2.79] | 1.77 [1.45 to 2.69]

5. Secondary Outcome: Phase 2: Objective Response Rate (ORR), as Assessed Using RECIST 1.1
Description: The ORR was defined as the percentage of participants with confirmed complete response (CR) or partial response (PR). CR: Disappearance of all target lesions and any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. Disappearance of all non-target lesions and normalisation of tumour marker level. All lymph nodes must be non-pathological in size (<10 mm short axis). PR: At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: From date of randomization to date of progression (maximum exposure: 24 cycles [each cycle = 14 days])
Population: FAS included all participants who were randomized in Phase 2 by following the intent-to-treat principle.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 2: Avelumab + Placebo | Phase 2: Avelumab + Entinostat
Number analyzed (Participants) | 41 | 85
percentage of participants | 4.88 [0.60 to 16.53] | 5.88 [1.94 to 13.20]

6. Secondary Outcome: Phase 2: ORR, as Assessed Using irRECIST
Description: The ORR was defined as the percentage of participants with confirmed CR or PR. CR: Complete disappearance of all lesions (whether measurable or not) and no new lesions. All measurable lymph nodes also must have a reduction in short axis to <10 mm. PR: Sum of the diameters (longest for non-nodal lesions, shortest for nodal lesions) of target and new measurable lesions decreases ≥30%.
Time Frame: From date of randomization to date of progression (maximum exposure: 24 cycles [each cycle = 14 days])
Population: FAS included all participants who were randomized in Phase 2 by following the intent-to-treat principle.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 2: Avelumab + Placebo | Phase 2: Avelumab + Entinostat
Number analyzed (Participants) | 41 | 85
percentage of participants | 2.44 [0.06 to 12.86] | 4.71 [1.30 to 11.61]

7. Secondary Outcome: Phase 2: Clinical Benefit Rate (CBR), as Assessed Using RECIST 1.1
Description: The CBR was defined as the percentage of participants with a confirmed CR, PR, or stable disease (SD) lasting for at least 6 months. CR: Disappearance of all target lesions and any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. Disappearance of all non-target lesions and normalisation of tumour marker level. All lymph nodes must be non-pathological in size (<10 mm short axis). PR: At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. SD: Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study.
Time Frame: From date of randomization to date of progression (maximum exposure: 24 cycles [each cycle = 14 days])
Population: FAS included all participants who were randomized in Phase 2 by following the intent-to-treat principle.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 2: Avelumab + Placebo | Phase 2: Avelumab + Entinostat
Number analyzed (Participants) | 41 | 85
percentage of participants | 9.76 [2.72 to 23.13] | 11.76 [5.79 to 20.57]

8. Secondary Outcome: Phase 2: CBR, as Assessed Using irRECIST
Description: The CBR was defined as the percentage of participants with a confirmed CR, PR, or SD lasting for at least 6 months. CR: Complete disappearance of all lesions (whether measurable or not) and no new lesions. All measurable lymph nodes also must have a reduction in short axis to <10 mm. PR: Sum of the diameters (longest for non-nodal lesions, shortest for nodal lesions) of target and new measurable lesions decreases ≥30%. SD: Sum of the diameters (longest for nonnodal lesions, shortest for nodal lesions) of target and new measurable lesions neither CR, PR, (compared to baseline) or PD (compared to nadir).
Time Frame: From date of randomization to date of progression (maximum exposure: 24 cycle [each cycle = 14 days])
Population: FAS included all participants who were randomized in Phase 2 by following the intent-to-treat principle.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 2: Avelumab + Placebo | Phase 2: Avelumab + Entinostat
Number analyzed (Participants) | 41 | 85
percentage of participants | 9.76 [2.72 to 23.13] | 9.41 [4.15 to 17.71]

9. Secondary Outcome: Phase 2: Overall Survival
Description: Overall survival was defined as the number of months from randomization to the date of death (due to any cause).
Time Frame: From date of randomization to the date of death (maximum exposure: 24 cycles [each cycle = 14 days])
Population: FAS included all participants who were randomized in Phase 2 by following the intent-to-treat principle.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 2: Avelumab + Placebo | Phase 2: Avelumab + Entinostat
Number analyzed (Participants) | 41 | 85
months | 10.55 [6.41 to 16.72] | 12.85 [9.53 to 18.37]

10. Secondary Outcome: Phase 2: Duration of Response
Description: Duration of response was defined as the number of months from the start date of PR or CR (whichever response occurred first) and subsequently confirmed, to the first date that recurrent or progressive disease was documented. CR: Disappearance of all target lesions and any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. Disappearance of all non-target lesions and normalisation of tumour marker level. All lymph nodes must be non-pathological in size (<10 mm short axis). PR: At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. PD: At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study .In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm; the appearance of one or more new lesions; and unequivocal progression of existing non-target lesions.
Time Frame: From start date of CR or PR to date of progression (maximum exposure: 24 cycles [each cycle = 14 days])
Population: FAS included all participants who were randomized in Phase 2 by following the intent-to-treat principle and had a response (achieved objective response: complete response or partial response).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 2: Avelumab + Placebo | Phase 2: Avelumab + Entinostat
Number analyzed (Participants) | 2 | 5
months | 6.83 [4.14 to NA] — Due to smaller number of participants with an event, upper limit of 95 % confidence interval (CI) could not be calculated. | 4.21 [2.17 to 16.59]

11. Secondary Outcome: Phase 2: Time to Response
Description: Time to response was defined as the number of months from the randomization date to the first date the participant achieved a PR or CR (whichever response occurred first and was subsequently confirmed). CR: Disappearance of all target lesions and any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. Disappearance of all non-target lesions and normalisation of tumour marker level. All lymph nodes must be non-pathological in size (<10 mm short axis). PR: At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: From the date of randomization to date of PR or CR (maximum exposure: 24 cycles [each cycle = 14 days])
Population: as for outcome 10
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 2: Avelumab + Placebo | Phase 2: Avelumab + Entinostat
Number analyzed (Participants) | 2 | 5
months | 2.10 [1.38 to 2.83] | 2.79 [1.35 to 4.17]

12. Secondary Outcome: Phase 1b: Number of Participants With Treatment-Emergent Adverse Events (TEAEs), Serious Adverse Events (SAEs), AEs Resulting in the Permanent Discontinuation of Study Drug, and Death
Description: An adverse event (AE) was defined as any untoward medical occurrence that develops or worsens in severity during the conduct of a clinical study and does not necessarily have a causal relationship to the study drug. SAEs included death, a life-threatening adverse event, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant disability or incapacity, a congenital anomaly or birth defect, or an important medical event that jeopardized the participant and required medical intervention to prevent 1 of the outcomes listed in this definition. TEAEs were defined as AEs that started on or after the first administration of study drug and within 30 days of the last administration of any study treatment. A summary of serious and non-serious AEs regardless of causality is located in 'Reported Adverse Events module'.
Time Frame: From first dose of study drug up to 30 days after end of treatment (maximum exposure: 24 cycles [each cycle = 14 days])
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1B: Avelumab + Entinostat (3 mg) | Phase 1B: Avelumab + Entinostat (5 mg)
Number analyzed (Participants) | 6 | 8
Participants
  Any TEAEs | 6 | 8
  Death | 1 | 0
  SAEs | 1 | 4
  AEs Resulting in the Permanent Discontinuation of Study Drug | 0 | 5

13. Secondary Outcome: Phase 2: Number of Participants With TEAEs, SAEs, AEs Resulting in the Permanent Discontinuation of Study Drug, and Death
Description: An AE was defined as any untoward medical occurrence that develops or worsens in severity during the conduct of a clinical study and does not necessarily have a causal relationship to the study drug. SAEs included death, a life-threatening adverse event, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant disability or incapacity, a congenital anomaly or birth defect, or an important medical event that jeopardized the participant and required medical intervention to prevent 1 of the outcomes listed in this definition. TEAEs were defined as AEs that started on or after the first administration of study drug and within 30 days of the last administration of any study treatment. A summary of serious and non-serious AEs regardless of causality is located in 'Reported Adverse Events module'.
Time Frame: From first dose of study drug up to 30 days after end of treatment (maximum exposure: 24 cycles [each cycle = 14 days])
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2: Avelumab + Placebo | Phase 2: Avelumab + Entinostat
Number analyzed (Participants) | 40 | 85
Participants
  Any TEAEs | 39 | 85
  Death | 1 | 1
  SAEs | 17 | 39
  AEs Resulting in the Permanent Discontinuation of Study Drug | 6 | 21

14. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero to Infinity (AUC0-inf) of Avelumab When Given in Combination With Entinostat
Time Frame: Pre-dose and post-infusion on Day 1 of Cycle 1 the 30-day follow-up (maximum exposure: 24 cycles [each cycle = 14 days])
Population: Analysis was not performed as data were not collected for this outcome measure.
Arm/Group | Phase 2: Avelumab + Entinostat
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to 30 days after end of treatment (maximum exposure: 24 cycles [each cycle = 14 days])
Description: Deaths were assessed for all participants enrolled in Phase 1b and randomized to treatment in Part 2. AEs were assessed for all participants who received at least 1 dose of either study drug, entinostat, or avelumab.
Arm/Group | Phase 1B: Avelumab + Entinostat (3 mg) | Phase 1B: Avelumab + Entinostat (5 mg) | Phase 2: Avelumab + Placebo | Phase 2: Avelumab + Entinostat
All-Cause Mortality (participants affected / at risk) | 5/6 | 4/8 | 26/41 | 54/85
Serious Adverse Events (participants affected / at risk) | 0/6 | 4/8 | 17/40 | 39/85
Other Adverse Events (participants affected / at risk) | 6/6 | 8/8 | 39/40 | 85/85
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1B: Avelumab + Entinostat (3 mg) (N=6) | Phase 1B: Avelumab + Entinostat (5 mg) (N=8) | Phase 2: Avelumab + Placebo (N=40) | Phase 2: Avelumab + Entinostat (N=85)
Paraneoplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Myasthenic syndrome (Nervous system disorders) | 0 | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Erosive oesophagitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 3 | 5
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 4
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 3
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 3
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 2
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 1 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 3
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 2 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 2
Asthenia (General disorders) | 0 | 0 | 0 | 2
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 0 | 2
Large intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Malignant ascites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 2
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 1
Bile duct obstruction (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 0 | 0 | 1
Cardiac failure congestive (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1
Cholangitis (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 0 | 1
Clostridium difficile infection (Infections and infestations) | 0 | 0 | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 1
Cystitis klebsiella (Infections and infestations) | 0 | 0 | 0 | 1
Device related infection (Infections and infestations) | 0 | 0 | 0 | 1
Device related sepsis (Infections and infestations) | 0 | 0 | 1 | 0
Disease progression (General disorders) | 0 | 0 | 0 | 1
Dysarthria (Nervous system disorders) | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Embolism (Vascular disorders) | 0 | 0 | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Infectious colitis (Infections and infestations) | 0 | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 0 | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Intestinal perforation (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Kidney infection (Infections and infestations) | 0 | 0 | 0 | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Necrotising fasciitis (Infections and infestations) | 0 | 0 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 1
Pericarditis (Cardiac disorders) | 0 | 0 | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Respiratory syncytial virus infection (Infections and infestations) | 0 | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 0 | 1
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Transaminases increased (Investigations) | 0 | 0 | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1B: Avelumab + Entinostat (3 mg) (N=6) | Phase 1B: Avelumab + Entinostat (5 mg) (N=8) | Phase 2: Avelumab + Placebo (N=40) | Phase 2: Avelumab + Entinostat (N=85)
Nausea (Gastrointestinal disorders) | 2 | 6 | 15 | 37
Diarrhoea (Gastrointestinal disorders) | 3 | 2 | 11 | 34
Abdominal pain (Gastrointestinal disorders) | 2 | 1 | 12 | 28
Vomiting (Gastrointestinal disorders) | 1 | 2 | 11 | 23
Constipation (Gastrointestinal disorders) | 0 | 4 | 11 | 24
Abdominal distension (Gastrointestinal disorders) | 3 | 1 | 5 | 9
Ascites (Gastrointestinal disorders) | 0 | 0 | 6 | 8
Dry mouth (Gastrointestinal disorders) | 1 | 1 | 6 | 8
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1 | 3 | 4
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 4 | 4
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 1 | 4 | 4
Anal incontinence (Gastrointestinal disorders) | 0 | 0 | 2 | 1
Flatulence (Gastrointestinal disorders) | 0 | 0 | 2 | 3
Fatigue (General disorders) | 2 | 6 | 17 | 51
Oedema peripheral (General disorders) | 1 | 1 | 3 | 24
Chills (General disorders) | 1 | 1 | 5 | 21
Pyrexia (General disorders) | 0 | 0 | 4 | 12
Asthenia (General disorders) | 0 | 1 | 4 | 2
Pain (General disorders) | 0 | 0 | 4 | 4
Influenza like illness (General disorders) | 0 | 0 | 2 | 5
Early satiety (General disorders) | 0 | 0 | 2 | 3
Malaise (General disorders) | 0 | 1 | 0 | 4
Decreased appetite (Metabolism and nutrition disorders) | 4 | 6 | 7 | 22
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 5 | 18
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 2 | 19
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1 | 3 | 14
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 3 | 9
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 11
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 14
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 7
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 4
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 7 | 20
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 8 | 17
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 8
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 5
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3 | 5
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 3 | 5
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 4 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 3 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 6 | 13
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 1 | 3 | 12
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 7 | 6
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 8
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 6
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3 | 3
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 4
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 9 | 24
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 16
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 11
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 4
Weight decreased (Investigations) | 0 | 2 | 5 | 8
Blood alkaline phosphatase increased (Investigations) | 1 | 0 | 1 | 10
Platelet count decreased (Investigations) | 1 | 1 | 0 | 11
Blood creatinine increased (Investigations) | 1 | 0 | 5 | 7
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 8
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 2 | 3
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 5
Headache (Nervous system disorders) | 1 | 2 | 8 | 11
Dizziness (Nervous system disorders) | 0 | 0 | 2 | 18
Dysgeusia (Nervous system disorders) | 0 | 1 | 0 | 5
Dysarthria (Nervous system disorders) | 0 | 0 | 2 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 4 | 8
Pneumonia (Infections and infestations) | 0 | 0 | 3 | 3
Upper respiratory tract infection (Infections and infestations) | 1 | 1 | 3 | 7
Skin infection (Infections and infestations) | 0 | 0 | 2 | 2
Rash (Skin and subcutaneous tissue disorders) | 1 | 1 | 3 | 7
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 4 | 5
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 5
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 3
Hypertension (Vascular disorders) | 0 | 2 | 4 | 7
Hypotension (Vascular disorders) | 0 | 0 | 2 | 6
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 1 | 4 | 6
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 3 | 6
Palpitations (Cardiac disorders) | 0 | 0 | 1 | 5
Tachycardia (Cardiac disorders) | 0 | 1 | 0 | 5
Anxiety (Psychiatric disorders) | 0 | 0 | 6 | 5
Insomnia (Psychiatric disorders) | 0 | 2 | 3 | 7
Depression (Psychiatric disorders) | 0 | 0 | 3 | 2
Dysuria (Renal and urinary disorders) | 0 | 2 | 2 | 4
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 2 | 2
Micturition urgency (Renal and urinary disorders) | 0 | 0 | 2 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 3 | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 3 | 0
Dry eye (Eye disorders) | 0 | 0 | 2 | 0
Hypothyroidism (Endocrine disorders) | 1 | 1 | 2 | 4
Malignant ascites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 1 | 1 | 3
Stomatitis (Gastrointestinal disorders) | 0 | 2 | 0 | 3
Diverticulum intestinal (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 1 | 0 | 2
Impaired gastric emptying (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gait disturbance (General disorders) | 0 | 1 | 1 | 0
Peripheral swelling (General disorders) | 1 | 0 | 0 | 4
Blood lactate dehydrogenase increased (Investigations) | 0 | 1 | 0 | 0
Breath sounds abnormal (Investigations) | 1 | 0 | 0 | 0
Weight increased (Investigations) | 1 | 0 | 0 | 2
Connective tissue disorder (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 3
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Myositis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Restless legs syndrome (Nervous system disorders) | 1 | 0 | 0 | 0
Flushing (Vascular disorders) | 1 | 0 | 0 | 1
Hot flush (Vascular disorders) | 0 | 1 | 0 | 2
Steroid withdrawal syndrome (Endocrine disorders) | 0 | 1 | 0 | 0
Pharyngitis (Infections and infestations) | 1 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 3
Scratch (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Mental status changes (Psychiatric disorders) | 0 | 1 | 0 | 1
Ear pain (Ear and labyrinth disorders) | 0 | 1 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publication of the results of the multi-center Study shall not be made before the first multi-site publication by Sponsor or Publications Committee. No Public Presentation by Institution or Investigator will be made until Study Documentation/Results from all sites are received and analyzed by Sponsor. Separate publication by Investigator will be delayed for a period of 18 months until the initial publication by Committee or Sponsor, or a determination is made not to make such publication.

DOCUMENTS (2):
  • Study Protocol (2017-02-02): https://cdn.clinicaltrials.gov/large-docs/23/NCT02915523/Prot_000.pdf
  • Statistical Analysis Plan (2018-07-24): https://cdn.clinicaltrials.gov/large-docs/23/NCT02915523/SAP_001.pdf